CLINICAL TRIAL: NCT04190732
Title: Impact of Physician Contact on Patient Anxiety and Distress During the Waiting Period After Embryo Transfer: a Randomized Controlled Study
Brief Title: Impact of Physician Contact on Patient Anxiety During the Waiting Period After Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boston IVF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019P000939
Record Dates: First submitted 2019-11-26; First posted 2019-12-09 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Infertility
Keywords: infertility; in-vitro fertilization (IVF); anxiety; distress
MeSH Terms: conditions — Infertility; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physician phone call (Experimental): Participants will receive a five-minute phone call from one physician 3 to 4 days after a fresh or frozen embryo transfer. The physician will not have access to patient specific IVF cycle details. The phone call will follow scripted questions and utilize scripted phrases to help minimize variation.
  Interventions: Behavioral: Physician phone call
- Routine care (No Intervention): Participants will receive routine care and no physician phone call will be performed during the waiting period between embryo transfer and the pregnancy test.

INTERVENTIONS:
Behavioral: Physician phone call — Often, patients will not have contact with a physician during the waiting period between embryo transfer and the pregnancy test. Participants in the intervention group will receive a phone call from one physician 3 to 4 days after fresh or frozen embryo transfer to check in. The physician will introduce themselves and state they are a part of the research team.
  Arms: Physician phone call

SUMMARY:
This will be a randomized controlled trial to compare if physician contact within the period from embryo transfer to serum pregnancy test decreases anxiety levels for first-time IVF patients.

DETAILED DESCRIPTION:
Overview This will be a randomized controlled trial to compare if physician contact within the period from embryo transfer to first pregnancy test decreases anxiety levels for first-time IVF patients.

Methods Study participation will not influence any element of IVF treatment, and all patients will be receiving the standard of care at Boston IVF. Potential participants will be identified by a member of the research team, who will review the appointment log and medical records to ensure eligibility. Participants who meet eligibility criteria will receive an email introduction to the study on the first stimulation day of the cycle and participants will be asked if interested in participating. Interested participants can click a secure REDCap link to learn more about that study. Participants who agree to participate will be directed via a unique link for each participant to a REDCap survey to complete a baseline questionnaire prior to the first ultrasound monitoring (T1), which is normally day 3 to 6 of IVF stimulation. Participants that complete the baseline survey are consenting for the study. Baseline demographic data will be obtained from the electronic medical record including: age, race, education level, partner status, height, weight, gravidity, and parity. Baseline clinical data, including anti-mullerian hormone and day 3 follicle stimulating hormone levels, will be obtained from the electronic medical record. The baseline survey will include demographic questions, the state-trait anxiety inventory (STAI), and the Hospital Anxiety and Depression Scale (HADS). STAI and HADS are two validated surveys used widely when examining anxiety in patients. The STAI is comprised of the trait and state questions. After stimulation day 3, a reminder email will be sent to eligible participants via REDCap to introduce the study again with a follow up phone call on stimulation day 4, if needed. Given the quick turnaround time from stimulation day 1 to first ultrasound monitoring (stimulation day 3 to 6), the additional email/phone contact schedule is necessary. If participants do not complete the baseline survey in entirety, participants will not be eligible for randomization. Participants will need to complete the survey in one sitting. Randomization will only occur if participants have an embryo transfer and complete the baseline survey. If selected to the intervention arm, participants will be called by one physician 3 to 4 days after the embryo transfer. Participants will be informed that the physician contact is not the participants specific doctor of record and that the physician contact will not be able to answer specific questions about the participants treatment cycle.

All participants that have an embryo transfer (fresh or frozen) will have a scheduled serum beta-hCG 10-12 days after the date of transfer. Eight days after the transfer (T2), participants will receive a second survey that will only include the STAI - state and HADS to be completed prior to the first serum beta-hCG. If participants have not started the survey by 9 days after the transfer, the participant will receive a reminder email on stimulation day 9 in the morning followed by a phone call on stimulation day 9 in the evening if needed for a reminder to complete the survey. The participant has the option to withdraw from the study at any time by notifying the research team by email or phone.

Intervention Participants will receive routine care or an approximately five-minute phone call from a physician 3 to 4 days after a fresh or frozen embryo transfer. The physician will state they are a part of the research team. For participants that do not answer the phone, a message will be left stating the participant will receive another phone call that same day and once more the following day if the participant does not answer on the second attempt. The phone call will follow scripted questions and utilize scripted phrases to help minimize variation.

Randomization Participants undergoing a fresh embryo transfer or planned frozen embryo transfer/PGT-A are eligible for inclusion in the study. Participants will be block-randomized by type of transfer to ensure balance between the intervention and control groups. The randomization scheme will be generated via REDCap. If participants are randomized to the intervention arm, participants will know this only if the participant receives a physician phone call during the waiting period after embryo transfers. All participants, regardless of transfer type, will be randomized only after participants have an embryo transfer.

Sample Size Justification The sample size calculation is based on data from a prior study that evaluated stress throughout the course of a IVF cycle using the STAI. The mean STAI-S in the infertility population ranges from 33-50, with Turner et al. reporting a mean STAI-S score of 40 ± 12. Assuming that the mean STAI-S score in the control group will be 40 ± 12 at the second time point, the investigators hypothesize that the mean STAI-S at this point in the intervention group will decrease to 35 ± 12. In order to achieve 80% power to detect the specified difference using a two-sided alpha of 0.05, the investigators will need 91 evaluable participants per arm. The Investigators anticipate that approximately 15% of participants will not complete the second survey, and the investigators will inflate the sample size by another 15% to account for a non-normal distribution. Thus, the investigators aim to randomize 121 participants per arm for a total of 242 participants.

Data Analysis Descriptive data will be presented as the proportion, mean with standard deviation, or median with interquartile range. Comparisons will be made using the chi-square or Fisher's exact test for categorical variables and parametric or non-parametric tests for continuous variables based on data distribution. All data will be analyzed with SAS 9.4 (SAS Institute Inc., Cary, NC, USA). All tests will be two sided and a P value <0.05 will be required to confer significance.

ELIGIBILITY:
Inclusion Criteria:

* First IVF cycle
* Autologous cycle
* 18 - 43 years of age

Exclusion Criteria:

* Utilizing a gestational carrier
* Preimplantation Genetic Testing for chromosome structural rearrangements (PGT- SR)
* Preimplantation Genetic Testing for Single gene (monogenic) (PGT-M)

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female patients undergoing In vitro fertilization treatment using their own eggs
Enrollment: 231 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety levels from two time points in an IVF cycle measured by the State Trait Anxiety Inventory - State (STAI-S) survey | Completed twice: once between IVF stimulation days 1-4 (T1) and again 8 days after (T2) embryo transfer and before first pregnancy test
  The investigators will assess change in anxiety levels from T1 to T2 using the State Trait Anxiety Inventory - State survey. A lower score on the State Trait Anxiety Inventory - State at T2 signifies a decrease in anxiety levels for a participant. The minimum and maximum score on the State Trait Anxiety Inventory - State is 20 and 80.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Penzias, MD, Principal Investigator — Boston IVF
Locations (1):
- Boston IVF, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No